CLINICAL TRIAL: NCT04049071
Title: Proposal for Establishment of a UK Post-marketing Surveillance Registry to Study the Effectiveness, Safety and Prescribing Habits of Tocilizumab for the Treatment of Giant Cell Arteritis in the UK National Health Service, Nested Within the Existing Structure of the UK GCA Consortium and UKIVAS Studies
Brief Title: TARGET GCAT Registry
Status: Terminated | Type: Observational
Why Stopped: Covid-19
Sponsor: University of Leeds (Other)
Collaborators: University of Oxford (Other); Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Ann Morgan, Professor of Molecular Rheumatology and Honorary Consultant Rheumatologist, University of Leeds
Other Study IDs: MM05/7307
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Giant Cell Arteritis
Keywords: Tocilizumab; Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Cases are patients that are prescribed tocilizumab as escalation therapy for relapsing/refractory GCA
- Control: Controls are those that are prescribed an alternative escalation therapy (not tocilizumab) for relapsing/refractory GCA.

SUMMARY:
A longitudinal post-marketing surveillance registry nested within the UK GCA Consortium that assesses the effectiveness and safety of tocilizumab in controlling refractory or relapsing forms of GCA in patients who require escalation of therapy to reach sustained remission. Half the patients recruited will have been prescribed tocilizumab (cases) and the other half will be prescribed alternative therapies (controls).

There are four study visits over 18 months: baseline, 6 months, 12 months and 18 months. At each visit data is collected on demographics; diagnosis and investigations; previous and concomitant medications; medical history; co-morbidities, vital signs; smoking and alcohol; disease activity and damage; routine laboratory tests; reason for starting escalation therapy. Safety data is collected on an ongoing basis.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a diagnosis of GCA and be eligible for the UK GCA Consortium study
* Willing and able to consent
* Have refractory or relapsing GCA as defined by the NHS England commissioning statement for tocilizumab.
* Require treatment escalation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 patients prescribed tocilizumab for GCA within the NHS and 500 age-, sex- and centre-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
To determine the proportion of eligible patients who achieve sustained partial or complete remission 6 months after the start of tocilizumab | 6 months
  Data on disease features and lab tests collected at 6 month, compared with that collected at baseline

SECONDARY OUTCOMES:
To determine the proportion of eligible patients who achieve a sustained complete remission 6 months after the start of tocilizumab | 6 months
  Data on disease features and lab tests collected at 6 month, compared with that collected at baseline
To assess the safety (event reporting) and effectiveness (in terms of prevention of relapse) of tocilizumab compared to other strategies for refractory/relapsing disease in patients with GCA who require escalation therapy. | 18 months
  Collection of safety data throughout study (non serious adverse events, serious adverse events, adverse events of special interest, special situations, notification of death)
To compare characteristics (demographics, disease severity, risk factors for steroid toxicity, contraindications to tocilizumab, concomitant medications) of real-world patients prescribed tocilizumab to clinical trial populations. | 0-18 months
  All data collected throughout the study period
To describe relapse rates in patients with GCA treated with tocilizumab at treatment completion (usually 12 months in the UK) and 6 months following discontinuation of tocilizumab | 0-18 months
  Data on disease features and lab tests collected at month 12 and 18 and compared with that collected at baseline and month 6
To describe disease activity during the first 6 and 12 months following the start of tocilizumab, compared to other treatment strategies for refractory/relapsing disease | 0-12 months
  Data collected on disease features, inflammatory markers and vital signs.
To describe ischaemic complications during the first 6 and 12 months following the start of tocilizumab, compared to other treatment strategies for refractory/relapsing disease | 0-12 months
  Data collected on disease features and event reporting as appropriate (serious adverse events & non-serious adverse events).
To describe drug related toxicity during the first 6 and 12 months following the start of tocilizumab, compared to other treatment strategies for refractory/relapsing disease | 0-12 months
  Data collected on lab results such as HbA1c and medication taken including the dose, reason for changes in dose or discontinuation, documentation of any events relating to drug toxicity.
To describe patterns of glucocorticoid dosing, including estimated cumulative dose & time to discontinuation of glucocorticoids, in patients with GCA & treated with tocilizumab, compared to other treatment strategies for refractory/relapsing disease | 0-18 months
  Data on glucocorticoid collected throughout study including dose changes & date of change
To describe reasons for premature discontinuation of tocilizumab | 0-18 months
  Reason for premature discontinuation of tocilizumab is captured at the follow up visits.
To estimate the prevalence of glucocorticoid toxicity (e.g. weight gain, fracture, diabetes, infection, or new psychiatric diagnosis) in patients with GCA who are treated with tocilizumab, compared to other strategies for refractory/relapsing disease | 0-18 months
  Data collected throughout study on features associated with glucocorticoid toxicity such as those listed within the title
To invite patients who agree to take part in the current study to consent to being approached to participate in future related studies of their condition, including randomised controlled trials | 0-18 months
  Keeping a record of those who have been agreed to be contacted for similar studies in the randomised controlled trials

CONTACTS AND LOCATIONS:
Overall Officials: Ann Morgan, Principal Investigator — University of Leeds
Locations (34):
- United Kingdom (34):
  - Birmingham Heartlands Hospital, Heart of England NHS Foundation Trust, Birmingham
  - Addenbrookes Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal Derby Hospital, University Hospital of Derby and Burton NHS Foundation Trust, Derby
  - Ninewells Hospital and Medical School, NHS Tayside, Dundee
  - NHS Lothian, Edinburgh, Edinburgh
  - Inverclyde Royal Hospital, NHS Greater Glasgow & Clyde, Glasgow
  - Royal Alexandra Hospital, NHS Greater Glasgow & Clyde, Glasgow
  - Vale of Leven Hospital, NHS Greater Glasgow & Clyde, Glasgow
  - Harrogate and District NHS Foundation Trust, Harrogate
  - Airedale General Hospital, Airedale NHS Foundation Trust, Keighley
  - Royal Lancaster & Westmorland General, University Hospitals of Morecambe Bay NHS Foundation Trust, Kendal
  - Chapel Allerton Hospital, Leeds Teaching Hospitals NHS Foundation Trust, Leeds
  - Leicester Royal Infirmary, University Hospitals of Leicester NHS Trust, Leicester
  - Aintree University Hospital, Aintree University Hospital NHS Foundation Trust, Liverpool
  - Royal Glamorgan Hospital, Cwm Taf University Health Board, Llantrisant
  - Kings College Hospital NHS Foundation Trust, London
  - Royal Free Hospital, Royal Free London NHS Foundation Trust, London
  - University College London NHS Foundation Trust, London
  - Luton and Dunstable Hospital, The Luton and Dunstable Hospitals NHS Foundation Trust, Luton
  - Manchester Royal Infirmary, Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - The Freeman Hospital, The Newcastle-upon-Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Northampton General Hospital, Northampton
  - Norfolk and Norwich University Hospital NHS Foundation Trust, Norwich
  - Queens Medical Centre, Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford Nuffield Orthopaedic Centre, Oxford University Hospitals NHS Foundation Trust, Oxford
  - Royal Preston Hospital, Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - Southend University Hospital NHS Foundation Trust, Southend-on-Sea
  - Lister Hospital, East and North Hertfordshire NHS Trust, Stevenage
  - Torbay Hospital, Torbay and South Devon NHS Foundation Trust, Torquay
  - Royal Cornwall Hospitals NHS Foundation Trust, Truro
  - Dewsbury & District Hospital, Mid Yorkshire Hospitals NHS Trust, Wakefield
  - Pinderfields Hospital, Mid Yorkshire Hospitals NHS Trust, Wakefield
  - University Hospital Wishaw, NHS Lanarkshire, Wishaw
  - York Teaching Hospital NHS Foundation Trust, York